CLINICAL TRIAL: NCT04567030
Title: Using Artificial Intelligence-platform on Plaque Control and Periodontal Treatment Outcome in Patients With Periodontal Disease-Preliminary Results
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-E(I)-20190141
Record Dates: First submitted 2020-09-24; First posted 2020-09-28 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Periodontal Diseases
Keywords: oral hygiene; artificial intelligence; Periodontitis; Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group A (AI Group: EG-A) (Experimental): Behavioral: AI intervention For the EG-A, a AI scan box will give to patients that taking mouth image at home once a week until six-month. The AI will send automated message to patients' mobile phone telling about their oral hygiene condition, gum condition, tooth condition.
  Interventions: Device: Dental monitoring (DM)
- Experimental group B (AI with humanized Group: EG-B) (Experimental): Behavioral: AI intervention For the EG-B,a AI scan box will give to patients that taking mouth image at home once a week until six-month. The AI will send automated message to patients' mobile phone telling about their oral hygiene condition, gum condition, tooth condition.
  The humanized counseling will also send to patients' mobile phone about each patients oral hygiene condition and advises.
  Interventions: Device: Dental monitoring (DM)
- Control group (CG) (No Intervention): the control group(CG) only have standard oral hygiene education

INTERVENTIONS:
Device: Dental monitoring (DM) — DM is the first APP system used in orthopedics patients in the world,it has been widely used in Asian countries (Taiwan, Hong Kong, Singapore, Japan, etc.) and has been used by 2140 patients so far. DM allows patients to take in-mouth photos at home, and uses AI as a background analysis to evaluate the patient's current oral condition (including oral hygiene and gum status) based on the photo.
  Arms: Experimental group A (AI Group: EG-A); Experimental group B (AI with humanized Group: EG-B)

SUMMARY:
The aim of this study was to evaluate the long-term effectiveness of an AI dental monitoring intervention on patients' periodontal disease, preventive behaviors and motivation. This randomized controlled trial included experimental group: AI group (EG-A), AI-humanized group (EG-B) and control group(CG), respectively.

The EG-A and EG-B received AI dental monitoring intervention by taking mouth image at home once a week for six month.

Baseline and follow-up surveys were used to collect the data in periodontal index, periodontal preventive behavior and motivation.

DETAILED DESCRIPTION:
A randomized experimental design was used. Patients with periodontal disease whose aged 35-65 years were recruited through department of Periodontics in Kaohsiung Medical University Hospital.

Each group was expected for 100 per group, patients will be randomized into each group. G*Power (version 3.1.9.4) was used for power analysis.

All patients will underwent periodontal examination at baseline and at 1-month, 3-month, 6-month follow-ups.

Each patients will be diagnosed periodontal disease by dentist and have more than 16 functional teeth.

Each patients will completed the questionnaire at baseline and at 1-month, 3-month and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35-65 years old
* Diagnosed periodontal disease by dentist (Comprehensive Periodontal Treatment Project)
* More than 16 functional teeth

Exclusion Criteria:

* Have received periodontal treatment within 3 months
* Patient has disease related to periodontal disease (ex. Drug-related excessive gum growth or blood clotting problems, pregnancy, mental illness)
* Disability patients

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
gingival index (GI) | Change from Baseline GI at 1-month after intervention
  The gingiva inflammation status of 6 tooth was recorded using the gingiva index, as follows:
  0 = No inflammation.
  1. = Mild inflammation, slight change in color, slight edema, no bleeding on probing
  2. = Moderate inflammation, moderate glazing, redness, bleeding on probing
  3. = Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
  For each patient, GI will measured by the teeth 12,16,24,32,36,44
gingival index (GI) | Change from Baseline GI at 3-month after intervention
  The gingiva inflammation status of 6 tooth was recorded using the gingiva index, as follows:
  0 = No inflammation.
  1. = Mild inflammation, slight change in color, slight edema, no bleeding on probing
  2. = Moderate inflammation, moderate glazing, redness, bleeding on probing
  3. = Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
  For each patient, GI will measured by the teeth 12,16,24,32,36,44
gingival index (GI) | Change from Baseline GI at 6-month after intervention
  The gingiva inflammation status of 6 tooth was recorded using the gingiva index, as follows:
  0 = No inflammation.
  1. = Mild inflammation, slight change in color, slight edema, no bleeding on probing
  2. = Moderate inflammation, moderate glazing, redness, bleeding on probing
  3. = Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
  For each patient, GI will measured by the teeth 12,16,24,32,36,44
plaque index (PI) | Change from Baseline PI at 1-month after intervention
  The plaque status of 6 tooth was recorded using the plaque index, as followes:
  0 = No plaque
  1. = Thin film of plaque, scraped with explorer
  2. = Moderate amount of plaque, visible with naked eyes
  3. = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  For each patient, PI will measured by the teeth 12,16,24,32,36,44
plaque index (PI) | Change from Baseline PI at 3-month after intervention
  The plaque status of 6 tooth was recorded using the plaque index, as followes:
  0 = No plaque
  1. = Thin film of plaque, scraped with explorer
  2. = Moderate amount of plaque, visible with naked eyes
  3. = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  For each patient, PI will measured by the teeth 12,16,24,32,36,44
plaque index (PI) | Change from Baseline PI at 6-month after intervention
  The plaque status of 6 tooth was recorded using the plaque index, as followes:
  0 = No plaque
  1. = Thin film of plaque, scraped with explorer
  2. = Moderate amount of plaque, visible with naked eyes
  3. = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  For each patient, PI will measured by the teeth 12,16,24,32,36,44
Probing Pocket Depth (PPD) | Change from Baseline PPD at 1-month after intervention
  Using periodontal probe to measure the depth from the bottom of the periodontal pocket to the gingival margin.
  For each patient, PPD will measured each teeth.
Probing Pocket Depth (PPD) | Change from Baseline PPD at 3-month after intervention
  Using periodontal probe to measure the depth from the bottom of the periodontal pocket to the gingival margin.
  For each patient, PPD will measured each teeth.
Probing Pocket Depth (PPD) | Change from Baseline PPD at 6-month after intervention
  Using periodontal probe to measure the depth from the bottom of the periodontal pocket to the gingival margin.
  For each patient, PPD will measured each teeth.
Clinical Attachment Loss(CAL) | Change from Baseline CAL at 1-month after intervention
  Using periodontal probe to measure the distance from the enamel-dentin junction to the bottom of the periodontal pocket.
  For each patient, CAL will measured each teeth.
Clinical Attachment Loss(CAL) | Change from Baseline CAL at 3-month after intervention
  Using periodontal probe to measure the distance from the enamel-dentin junction to the bottom of the periodontal pocket.
  For each patient, CAL will measured each teeth.
Clinical Attachment Loss(CAL) | Change from Baseline CAL at 6-month after intervention
  Using periodontal probe to measure the distance from the enamel-dentin junction to the bottom of the periodontal pocket.
  For each patient, CAL will measured each teeth.
Protection Motivation Theory (PMT) scores | Change from Baseline PMT at 1-month after intervention
  Item including that "I think periodontal disease is a serious disease" "If I do not have periodontal disease prevention behavior, the risk of developing periodontal disease in the future is very high" "If I stick to periodontal disease prevention behavior, it will improve my oral health" "I believe that I can follow the periodontal health guidance" "I find it hard to remember/hard to do periodontal health care guidance" "Periodontal disease bothers me" "I want to complete my personal periodontal disease prevention behavior plan" All the items' scores ranged from one to ten, with higher scores indicating a higher level of motivation toward change behaviors.
  Cronbach's α was 0.70 for this scale.The scores ranged from one ("impossible") to ten ("very possible"), with the total possible score ranging from seven to seventy.
Protection Motivation Theory (PMT) scores | Change from Baseline PMT at 3-month after intervention
  Item including that "I think periodontal disease is a serious disease" "If I do not have periodontal disease prevention behavior, the risk of developing periodontal disease in the future is very high" "If I stick to periodontal disease prevention behavior, it will improve my oral health" "I believe that I can follow the periodontal health guidance" "I find it hard to remember/hard to do periodontal health care guidance" "Periodontal disease bothers me" "I want to complete my personal periodontal disease prevention behavior plan" All the items' scores ranged from one to ten, with higher scores indicating a higher level of motivation toward change behaviors.
  Cronbach's α was 0.70 for this scale.The scores ranged from one ("impossible") to ten ("very possible"), with the total possible score ranging from seven to seventy.
Protection Motivation Theory (PMT) scores | Change from Baseline PMT at 6-month after intervention
  Item including that "I think periodontal disease is a serious disease" "If I do not have periodontal disease prevention behavior, the risk of developing periodontal disease in the future is very high" "If I stick to periodontal disease prevention behavior, it will improve my oral health" "I believe that I can follow the periodontal health guidance" "I find it hard to remember/hard to do periodontal health care guidance" "Periodontal disease bothers me" "I want to complete my personal periodontal disease prevention behavior plan" All the items' scores ranged from one to ten, with higher scores indicating a higher level of motivation toward change behaviors.
  Cronbach's α was 0.70 for this scale. The scores ranged from one ("impossible") to ten ("very possible"), with the total possible score ranging from seven to seventy.

SECONDARY OUTCOMES:
oral self-care behavior | Change from Baseline at 1 month after intervention
  Item including that "How many times do you brush your teeth a day?" The response was (once or twice day or three times or fours times or more/ day).
  "How long do you usually brush your teeth each time?" The response was lower than 1 min or 1-2 min or 2-3 min or more than 3 min/ day.
  "What is your main method of brushing your teeth?"The response was horizontally or vertically or Circle brush or Rotating brush or Horizontal+vertical+ and by the gum at a 45 degree angle. "How often do you replace your toothbrush?" The response was 3-6 month or more than 6 month or lower than 1 month or 1-2 month or 2-3 month.
  "Do you use a soft-bristled toothbrush?" The response was no or unknown or yes. "Do you have a habit of using interdental brushes?" The response was no or yes. "Do you have a habit of eating snack?" The response was no or yes.
oral self-care behavior | Change from Baseline at 3 month after intervention
  Item including that "How many times do you brush your teeth a day?" The response was (once or twice day or three times or fours times or more/ day).
  "How long do you usually brush your teeth each time?" The response was lower than 1 min or 1-2 min or 2-3 min or more than 3 min/ day.
  "What is your main method of brushing your teeth?"The response was horizontally or vertically or Circle brush or Rotating brush or Horizontal+vertical+ and by the gum at a 45 degree angle. "How often do you replace your toothbrush?" The response was 3-6 month or more than 6 month or lower than 1 month or 1-2 month or 2-3 month.
  "Do you use a soft-bristled toothbrush?" The response was no or unknown or yes. "Do you have a habit of using interdental brushes?" The response was no or yes. "Do you have a habit of eating snack?" The response was no or yes.
oral self-care behavior | Change from Baseline at 6 month after intervention
  Item including that "How many times do you brush your teeth a day?" The response was (once or twice day or three times or fours times or more/ day).
  "How long do you usually brush your teeth each time?" The response was lower than 1 min or 1-2 min or 2-3 min or more than 3 min/ day.
  "What is your main method of brushing your teeth?"The response was horizontally or vertically or Circle brush or Rotating brush or Horizontal+vertical+ and by the gum at a 45 degree angle. "How often do you replace your toothbrush?" The response was 3-6 month or more than 6 month or lower than 1 month or 1-2 month or 2-3 month.
  "Do you use a soft-bristled toothbrush?" The response was no or unknown or yes. "Do you have a habit of using interdental brushes?" The response was no or yes. "Do you have a habit of eating snack?" The response was no or yes.
OHIP-14T scales | Change from Baseline at 1 month after intervention
  Item including that because of problems with your teeth or mouth, you:
  "Have you had trouble pronouncing any words because of problems" "Have you felt that your sense of taste has worsened" "Have you had painful aching in your mouth" "Have you found it uncomfortable to eat any foods" "Have you been self-conscious" "Have you felt tense" "Has been your diet been unsatisfactory" "Have you had to interrupt meals?" "Have you found it difficult to relax" "Have you been a bit embarrassed" "Have you been a bit irritable with other people" "Have you had difficulty doing your usual jobs" "Have you felt that life in general was less satisfying" "Have you been totally unable to function" The scores ranged from one ("never") to five ("always"), with the total possible score ranging from fourteen to seventy.
OHIP-14T scales | Change from Baseline at 3 month after intervention
  Item including that because of problems with your teeth or mouth, you:
  "Have you had trouble pronouncing any words because of problems" "Have you felt that your sense of taste has worsened" "Have you had painful aching in your mouth" "Have you found it uncomfortable to eat any foods" "Have you been self-conscious" "Have you felt tense" "Has been your diet been unsatisfactory" "Have you had to interrupt meals?" "Have you found it difficult to relax" "Have you been a bit embarrassed" "Have you been a bit irritable with other people" "Have you had difficulty doing your usual jobs" "Have you felt that life in general was less satisfying" "Have you been totally unable to function" The scores ranged from one ("never") to five ("always"), with the total possible score ranging from fourteen to seventy.
OHIP-14T scales | Change from Baseline at 6 month after intervention
  Item including that because of problems with your teeth or mouth, you:
  "Have you had trouble pronouncing any words because of problems" "Have you felt that your sense of taste has worsened" "Have you had painful aching in your mouth" "Have you found it uncomfortable to eat any foods" "Have you been self-conscious" "Have you felt tense" "Has been your diet been unsatisfactory" "Have you had to interrupt meals?" "Have you found it difficult to relax" "Have you been a bit embarrassed" "Have you been a bit irritable with other people" "Have you had difficulty doing your usual jobs" "Have you felt that life in general was less satisfying" "Have you been totally unable to function" The scores ranged from one ("never") to five ("always"), with the total possible score ranging from fourteen to seventy.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Shen KL, Huang CL, Lin YC, Du JK, Chen FL, Kabasawa Y, Chen CC, Huang HL. Effects of artificial intelligence-assisted dental monitoring intervention in patients with periodontitis: A randomized controlled trial. J Clin Periodontol. 2022 Oct;49(10):988-998. doi: 10.1111/jcpe.13675. Epub 2022 Jul 10. PMID 35713224